CLINICAL TRIAL: NCT05292066
Title: Efficacy of Variable Doses of Pregabalin Vs Duloxetine in Diabetic Peripheral Neuropathic Pain: A Comparative Study
Brief Title: Efficacy of Pregabalin Vs Duloxetine in Diabetic Peripheral Neuropathic Pain at Variable Dose
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, NASEER AHMED, Fahim Ullah, Assistant professor., Rehman Medical Institute - RMI
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 07124
Record Dates: First submitted 2022-02-09; First posted 2022-03-23 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Diabetic Peripheral Neuropathic Pain
MeSH Terms: interventions — Duloxetine Hydrochloride; Pregabalin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Duloxetine Group (Other): Oral intake Duloxetine tablets, 30mg/day for 12 weeks.
  Interventions: Drug: Duloxetine Tablets,
- Pregabalin Group (Other): Oral intake of Pregabalin tablets, 75 mg/day for 12 weeks.
  Interventions: Drug: Pregabalin Tablets

INTERVENTIONS:
Drug: Duloxetine Tablets, — Duloxetine is an FDA-approved medication used to treat the major depressive disorder, generalized anxiety disorder, fibromyalgia, and neuropathic pain. It is taken by mouth. It is a serotonin-norepinephrine reuptake inhibitor.
  Pregabalin is an FDA approved, sold under the brand name Lyrica. it is an anticonvulsant and anxiolytic medication used to treat epilepsy, neuropathic pain, fibromyalgia, restless leg syndrome,
  Other Names: Cymbalta,
  Arms: Duloxetine Group
Drug: Pregabalin Tablets — Pregabalin is an FDA approved, it is an anticonvulsant and anxiolytic medication used to treat epilepsy, neuropathic pain, fibromyalgia, restless leg syndrome,
  Other Names: Lyrica.
  Arms: Pregabalin Group

SUMMARY:
Background Diabetic neuropathy is a widespread, debilitating condition and its management needs a significant cost. Around, 50% of diabetes mellitus (DM) patients suffer from Diabetic Peripheral Neuropathic Pain (DPNP). According to the reported data, specific anticonvulsants and antidepressants are effective for coping diabetic peripheral neuropathy. Two drugs, duloxetine and pregabalin, are officially permitted by the Food and Drug Administration (FDA) for the management of DPNP.

Methodology A Prospective Randomized Controlled Trial (RCT) trial for 12 weeks will be carried out on 126 volunteer DPNP patients with age between 18- to 70-year-old and participants was selected through consecutive sampling and will be evaluated on the basis of duration of the disease, pain scales and the data provided by particular consultants. The parameters will be measured weekly and final parameters will be measured after 12 weeks. Statistical analysis will be carried out by SPSS, ANOVA, and t-test.

Expected outcomes:

From this experimental design, investigators are expecting improvement in the management of DPNP and Duloxetine is more effective for treating patients suffering from DPNP.

DETAILED DESCRIPTION:
This is prospective clinical research, that will be executed from Feb 2022 to May 2022, including, only those patients who are diagnosed with DPNP of at least six months duration, attending Rehman Medical Institute, General hospital. The diagnosis will be primarily clinical.

Randomization of participants will be accomplished by registering the patients into any of two groups (Duloxetine group A, Pregabalin group B) using a statistical computer program. In group A (Duloxetine group) patients will receive duloxetine 30mg/day and group B (Pregabalin group) will receive Pregabalin 75 mg/day for upto 12 weeks.

Biothesiometry will be performed for all diagnosed diabetic patients. Relevant clinical tests like HBA1c, Lipid profile, TSH, vitamin B12 levels will be performed in all patients before randomization.

The sample size was calculated using an open epi sample size calculator using confidence interval 95%, power 80.

Mean ±SD of Duloxetine group was 5.60 ±0.89. Mean ±SD of Pregabalin group was 6.01±0.82. Pregabalin group sample size was calculated to be 63 patients, Duloxetine group sample size was calculated to be 63 patients. Total number of participants was 126.

Only, the approved procedures and protocols will be followed and all patients provided informed consent.

Demographic profiles of volunteer participants like age, gender, living arrangements and others will be noted down. History of disease like duration and treatment for diabetes will be documented. Biothesiometer score above 15 volts will be considered as DNPN. Relevant investigations like HBA1c, Lipid profile, TSH, vitamin B12 levels will be performed in all patients before randomization.

The criteria of classification for DPN will be done on the basis of the proposed TCSS score: zero to five points, without DPN; six to eight points, mild DPN; nine to 11 points, moderate DPN; and 12 to 19 points, severe DPN. The TCSS will be employed in people with type 2 diabetes to assess the prevalence of painful DPNP. A questionnaire (DN-4) will be used to evaluate the pain extent and the adverse effects related to duloxetine and pregabalin will be recorded in all cases.

Toronto clinical neuropathy score (TCNS), consists of three parts: symptom scores, reflex scores, and sensory test scores. The maximum score is 19 points. Better pain relief will be the primary outcome of the proposed study which will be evaluated as a decrease in visual analogue scale (VAS) score.

Written informed consent will be taken from each participant. Patients will be included in the study after informed consent and the patients have the right to withdraw from the trial at any point they want.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female patient with age more than 18 years to 70 years.
* Patients diagnosed with peripheral neuropathic pain affected by diabetes from at least 24 weeks and all other causes off peripheral painful neuropathy has been already excluded by their primary physician.
* Patients who may agree with written inform consent.
* HbA1c ≥ 6.5% and ≤ 10%

Exclusion Criteria:

* Patients with severe hepatic disease, cardiovascular diseases, Epilepsy and respiratory diseases or any other medical or psychiatric disorders.
* Patients with uncontrolled hypertension.
* DM patients with foot ulcers, foot injuries or any other painful lesion.
* Patients who are already using or used duloxetine or pregabalin in last three month.
* Pregnant women or those who may not agree to use medical recommended birth control procedures during the treatment.
* Patient with thyroid known disorders or diagnosed during the screening
* Vitamin B12 deficient patient
* Chronic alcoholics
* DKD, with eGFR < 30ml/min
* Hypertriglycedmia (TGs more then 250mg/dl)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
visual analogue scale score. | 3 months.
  Evaluation perceived pain intensity by patients
Toronto clinical neuropathy score | 3 months.
  Final diagnosis and staging of diabetic peripheral neuropathy of patients.
  Diabetes severity will be graded according to the results of this score.
  Out of a total score of 19, the grades are defined as follows:
  0-5 = no neuropathy; 6-8 = mild neuropathy; 9-11 = moderate neuropathy;
  ≥ 12 = severe neuropathy.

IPD SHARING:
Plan to Share IPD: Undecided